CLINICAL TRIAL: NCT03473743
Title: A Phase 1b-2 Study to Evaluate Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Various Regimens of Erdafitinib in Subjects With Metastatic or Locally Advanced Urothelial Cancer
Brief Title: A Study of Erdafitinib in Participants With Metastatic or Locally Advanced Urothelial Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108445; 42756493BLC2002 (Other: Janssen Research & Development, LLC); 2017-001980-19 (EudraCT Number); 2023-510295-31-00 (Registry Identifier: EUCT number)
Expanded Access: NCT03825484 (Approved for marketing)
Record Dates: First submitted 2018-03-14; First posted 2018-03-22 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — erdafitinib; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b: Dose Escalation (Experimental): Two dosing cohorts (erdafitinib and cetrelimab; and erdafitinib, cetrelimab and cisplatin/carboplatin) are explored in Phase 1b of the study. Participants will receive erdafitinib orally followed by cetrelimab intravenously (IV) and carboplatin/cisplatin IV as a part of platinum chemotherapy. The dose levels will be escalated sequentially based on the decisions of the Study Evaluation Team (SET) until the recommended Phase 2 Dose (RP2D) has been identified.
  Interventions: Drug: Erdafitinib; Drug: Cetrelimab; Drug: Cisplatin; Drug: Carboplatin
- Phase 2: Dose Expansion (Experimental): The participants will be randomized in a 1:1 manner to receive either erdafitinib alone (orally) or the identified RP2D of Phase 1b for erdafitinib (orally) in combination with cetrelimab (IV).
  Interventions: Drug: Erdafitinib; Drug: Cetrelimab

INTERVENTIONS:
Drug: Erdafitinib — Participants will receive erdafitinib orally.
  Other Names: JNJ-42756493
Drug: Cetrelimab — Participants will receive cetrelimab by intravenous infusion.
  Other Names: JNJ-63723283
Drug: Cisplatin — Participants will receive cisplatin by intravenous infusion as a part of platinum chemotherapy.
  Arms: Phase 1b: Dose Escalation
Drug: Carboplatin — Participants will receive carboplatin by intravenous infusion as a part of platinum chemotherapy.
  Arms: Phase 1b: Dose Escalation

SUMMARY:
The purpose of this study is to: (a) characterize the safety and tolerability of and to identify the recommended Phase 2 dose (RP2D) and schedule for erdafitinib in combination with cetrelimab, and for erdafitinib in combination with cetrelimab and platinum (cisplatin and carboplatin) chemotherapy and; (b) to evaluate the safety and clinical activity of erdafitinib alone and in combination with cetrelimab in cisplatin-ineligible participants with metastatic or locally advanced urothelial cancer (UC) with select fibroblast growth factor receptor (FGFR) gene alterations and no prior systemic therapy for metastatic disease.

DETAILED DESCRIPTION:
This open-label (all people know identity of intervention) and multicenter (when more than one hospital or medical school team work on a medical research study) study to establish the recommended phase 2 dose (RP2D) for erdafitinib and cetrelimab and/or platinum (cisplatin or carboplatin) chemotherapy, and to evaluate the safety of erdafitinib in combination with cetrelimab and platinum chemotherapy in Phase 1b and to evaluate the safety and efficacy of the RP2D of erdafitinib plus cetrelimab versus erdafitinib in Phase 2 in participants with advanced urothelial cancer with select fibroblast growth factor receptor (FGFR) gene alterations. Participants enrolled in Phase 1b erdafitinib + cetrelimab cohort may have received any number of lines of prior therapy, and participants enrolled in Phase 1b erdafitinib + cetrelimab + platinum chemotherapy cohort will have had no prior systemic therapy for metastatic disease and participants enrolled in Phase 2 will have had no prior systemic therapy for metastatic disease and will be cis-ineligible. Part 1 (Phase 1b: Dose Escalation) will identify safety and RP2Ds of erdafitinib + cetrelimab and erdafitinib + cetrelimab + platinum (cisplatin or carboplatin) chemotherapy, and Part 2 (Phase 2: Dose Expansion) will evaluate erdafitinib monotherapy and the RP2D regimen of the erdafitinib + cetrelimab combination to further characterize safety and clinical activity. The study will be conducted in 3 phases: screening phase, treatment phase, and follow-up phase. Study evaluations include efficacy, pharmacokinetics, pharmacodynamics, immunogenicity, biomarkers, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Histologic demonstration of transitional cell carcinoma of the urothelium. Variant urothelial carcinoma histologies such as glandular or squamous differentiation, or evolution to more aggressive phenotypes such as sarcomatoid or micropapillary change are acceptable
* Metastatic or locally advanced urothelial cancer
* Must have measurable disease by radiological imaging according to the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) at baseline
* Prior systemic therapy for metastatic urothelial cancer: (a) For Phase 1b erdafitinib + cetrelimab cohort: Any number of lines of prior therapy; (b) For Phase 1b erdafitinib + cetrelimab + platinum chemotherapy cohort: No prior systemic therapy for metastatic disease; and renal function for participants must have a creatinine clearance (CrCl) greater than (>) 30 milliliter per minute (mL/min) to receive carboplatin and >60 mL/min to receive cisplatin as calculated by Cockcroft Gault and (c) Phase 2: No prior systemic therapy for metastatic disease and cisplatin-ineligible based on: ECOG PS 0-1 and at least one of the following criteria: Renal function defined as creatinine clearance (CrCl) less than (˂) 60 mL/min as calculated by Cockcroft-Gault; Grade 2 or higher peripheral neuropathy per NCI-CTCAE version 5.0; Grade 2 or higher hearing loss per NCI-CTCAE version 5.0 OR ECOG PS 2
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) grade of: (a) Phase 1b erdafitinib + cetrelimab cohort: ECOG 0-2; (b) Phase 1b erdafitinib + cetrelimab + platinum chemotherapy cohort: ECOG 0-1 for cisplatin and 0-2 for carboplatin (c) Phase 2: ECOG 0-2

Exclusion Criteria:

* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 30 days prior to Cycle 1 Day 1. For Phase 1b, participants who have received the following prior antitumor therapy: received nitrosoureas and mitomycin C within 6 weeks
* Phase 1b erdafitinib + cetrelimab cohort: Chemotherapy within 3 weeks of Cycle 1 Day 1; Phase 1b erdafitinib + cetrelimab + platinum chemotherapy cohort and Phase 2: Prior neoadjuvant/adjuvant chemotherapy is allowed if the last dose was given >12 months prior to recurrent disease progression and did not result in drug-related toxicity leading to treatment discontinuation
* Prior anti-programmed death receptor-1 (PD-1), anti-programmed death ligand-1 (PD-L1), or anti-programmed death ligand-2 (PD-L2) therapy. Prior neoadjuvant/adjuvant checkpoint inhibitor therapy is allowed if the last dose was given more than (>)12 months prior to recurrent disease progression and did not result in drug-related toxicity leading to treatment discontinuation. PD-1 for non-muscle invasive bladder cancer is also allowed
* Active malignancies requiring concurrent therapy other than urothelial cancer
* Symptomatic central nervous system metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (127):
- United States (12):
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Norton Cancer Institute, Louisville, Kentucky
  - Maryland Oncology Hematology, PA, Rockville, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College - NY Presbyterian Hospital, New York, New York
  - White Plains Hospital Center for Cancer Care, White Plains, New York
  - Levine Cancer Institute, Carolinas HealthCare System, Charlotte, North Carolina
  - Toledo Clinic Cancer Centers, Toledo, Ohio
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Texas Oncology, P.A., Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Belarus (7):
  - Brest Regional Oncology Dispensary, Brest
  - Grodno University Hospital, Grodno
  - Gomel Regional Clinical Oncology Dispensary, Homyel
  - State Institution N.N. Alexandrov Republican Scientific and, Lesnoy
  - Minsk city Clinical Oncological Dispensary, Minsk
  - Mogilev Regional Hospital, Mogilev
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Belgium (7):
  - ULB Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Jolimont, Haine-Saint-Paul
  - Az Groeninge, Kortrijk
  - CHU de Liège - Domaine Universitaire du Sart Tilman, Liège
  - AZ Nikolaas - Campus Sint-Niklaas Moerland, Sint-Niklaas
  - GZA Ziekenhuizen- Campus St Augustinus, Wilrijk
- Brazil (7):
  - Fundacao Pio XII, Barretos
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Oncocentro Servicos Medicos e Hospitalares Ltda - Oncocentro, Fortaleza
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - CEPHO Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
- France (11):
  - Institut de Cancerologie de Ouest (ICO) Site Paul Papin, Angers
  - Hopital Saint André, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre hospitalier Saint Louis, La Rochelle
  - Centre Leon Berard, Lyon
  - APHM Hopital Timone, Marseille
  - Hopital Europeen Georges Pompidou, Paris
  - Clinique Sainte Anne, Strasbourg
  - CHRU de Tours, Tours
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Italy (15):
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Istituto di Candiolo, IRCCS, Candiolo
  - Ospedale Di Zona B Ramazzini, Carpi
  - UOS Oncologia Medica, A.O. Cannizzaro, Catania
  - Arcispedale S. Anna Ferrara, Ferrara
  - PO A.Manzoni di Lecco, ASST Lecco - Oncologia Medica - Lecco, Lecco
  - Ospedale Civile Di Livorno, Livorno
  - IRCCS Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale S. Maria Della Misericordia Centro Operativo Studi Clinici SC Oncologia Medica, Perugia
  - AUSL DI PIACENZA - Ospedale Guglielmo da Saliceto, Piacenza
  - Campus Bio Medico di Roma, Roma
  - Azienda Socio Sanitaria Territoriale (ASST) della Valtellin, Sondrio
  - Azienda Ospedaliera S. Maria Terni, Terni
  - Azienda Ospedaliero Universitaria S.Maria Della Misericordia, Udine
- Poland (4):
  - Przychodnia Lekarska KOMED Roman Karaszewski, Konin
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im M Kopernika w Lodzi, Lodz
  - LUX MED Onkologia Sp. z o.o., Warsaw
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
- Russia (15):
  - Altai Regional Oncology Dispensary, Barnaul
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - GUZ Kursk Regional Oncology Dispensary, Kislino Village
  - Leningrad Regional Oncology Dispensary, Kuzmolovsky
  - City Clinical Hospital n.a. D.D.Pletnev, Moscow
  - Russian Scientific Center of Roentgenoradiology, Moscow
  - Moscow City Clinical Hospital # 62, Moscow
  - Clinical Diagnostic Centre of Nizhny Novgorod Region, Nizhny Novgorod
  - Privolzhsky District Medical Centre, Nizhny Novgorod
  - Clinical Oncology Dispensary, Omsk
  - LLC Novaya Clinica, Pyatigorsk
  - Private Medical Institution Euromedservice, Saint Petersburg
  - Russian Scientific Center of Radiology and Surgical Technologies, Saint Petersburg
  - Tambov Regional Oncology Clinical Dispansary, Tambov
  - Multifunctional clinical medical center 'Medical city', Tyumen
- South Korea (10):
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - The Catholic university of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (17):
  - Hosp. Del Mar, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Complexo Hosp. Univ. de Ourense, Ourense
  - Complejo Hospitalario de Vigo, Pontevedra
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. Marques de Valdecilla, Santander
  - H. Clinico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. Virgen Del Rocio, Seville
  - Instituto Valenciano de Oncologia, Valencia
  - Hosp. Clinico Univ. de Valencia, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- Turkey (Türkiye) (12):
  - Adana Acibadem Hospital, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Adnan Menderes University Training and Research Hospital, Aydin
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Istanbul Medeniyet University Goztepe Training and Research Hospital, Istanbul
  - Ege University, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Karadeniz Teknik University Medical Faculty, Trabzon
- United Kingdom (4):
  - Royal Lancaster Infirmary, Lancaster
  - St Bartholomew's Hospital, London
  - University College London Hospitals Nhs Foundation Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- [Derived] LaRoche JK, Lanier J, Alvarenga R, Collins M, Costelloe T, Chiau A, Whetherly H, De Soete W, Faludi J, Rens K. Climate footprint of industry-sponsored in-human clinical trials: life cycle assessments of clinical trials spanning multiple phases and disease areas. BMJ Open. 2025 Feb 19;15(2):e085364. doi: 10.1136/bmjopen-2024-085364. PMID 39971605

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort Dose Level (DL) 1 (Phase 1b): Erdafitinib 6 Milligrams (mg) + Cetrelimab 240/480 mg: Participants received an oral tablet of erdafitinib 6 mg once daily in 28-day cycle starting from Cycle 1 Day 1 followed by intravenous (IV) injection of cetrelimab 240 mg every 2 weeks in 28-day cycle starting from Cycle 1 Day 1 up to Cycle 4 Day 15. From Cycle 5 Day 1, all participants received an increased dose of cetrelimab 480 mg every 4 weeks in 28-day cycle until disease progression, unacceptable toxicity (based on investigator assessment), or another treatment discontinuation criterion was met.
- Cohort DL2A (Phase 1b): Erdafitinib 8 mg + Cetrelimab 240/480 mg; Arm B (Phase 2): Erdafitinib 8 mg + Cetrelimab 240/480 mg: Participants received an oral tablet of erdafitinib 8 mg once daily in 28-day cycle starting from Cycle 1 Day 1 followed by IV injection of cetrelimab 240 mg every 2 weeks in 28-day cycle starting from Cycle 1 Day 1 up to Cycle 4 Day 15. From Cycle 5 Day 1, all participants received an increased dose of cetrelimab 480 mg every 4 weeks in 28-day cycle until disease progression, unacceptable toxicity (based on investigator assessment), or another treatment discontinuation criterion was met..
- Cohort DL2B (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg: Participants received an oral tablet of erdafitinib 8 mg once daily in 28-day cycle starting from Cycle 1 Day 1 followed by IV injection of cetrelimab 240 mg every 2 weeks in 28-day cycle starting from Cycle 2 Day 1 up to Cycle 4 Day 15. Based on phosphate (PO4) levels, erdafitinib dose was up-titrated to 9 mg once daily starting from Cycle 1 Day 15. From Cycle 5 Day 1, all participants received an increased dose of cetrelimab 480 mg every 4 weeks in 28-day cycle until disease progression, unacceptable toxicity (based on investigator assessment), or another treatment discontinuation criterion was met.
- Cohort DL2 (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg (RP2D): Participants received an oral tablet of recommended Phase 2 dose (RP2D) of erdafitinib 8 mg once daily in 28-day cycle starting from Cycle 1 Day 1 followed by IV injection of cetrelimab 240 mg every 2 weeks in 28-day cycle starting from Cycle 1 Day 1 up to Cycle 4 Day 15. Based on PO4 levels, erdafitinib dose was up-titrated to 9 mg, orally, once daily starting from Cycle 1 Day 15. From Cycle 5 Day 1, all participants received an increased dose of cetrelimab 480 mg every 4 weeks in 28-day cycle until disease progression, unacceptable toxicity (based on investigator assessment), or another treatment discontinuation criterion was met.
- Cohort DL2C (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Cisplatin 50 mg/m^2: Participants received an oral tablet of erdafitinib 8 mg once daily in 28-day cycle starting from Cycle 1 Day 1 along with single dose of IV injection of cetrelimab 360 mg and cisplatin 50 milligrams per meter square (mg/m^2) (chemotherapy) every 2 weeks in 28-day cycle starting from Cycle 1 Day 1 until disease progression, unacceptable toxicity (based on investigator assessment), or another treatment discontinuation criterion was met.
- Cohort DL2D (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Carboplatin AUC 4 mg/mL/Min: Participants received an oral tablet of erdafitinib 8 mg once daily in 28-day cycle starting from Cycle 1 Day 1 along with single dose of IV injection of cetrelimab 360 mg and carboplatin area under the curve (AUC) 4 milligrams per milliliter per minute (mg/mL/min) (chemotherapy) every 2 weeks in 28-day cycle starting from Cycle 1 Day 1 until disease progression, unacceptable toxicity (based on investigator assessment), or another treatment discontinuation criterion was met.
- Arm A (Phase 2): Erdafitinib 8/9 mg Monotherapy: Participants received an oral tablet of erdafitinib 8 mg once daily in 28-day cycle starting from Cycle 1 Day 1. Based on PO4 levels, erdafitinib dose was up-titrated to 9 mg, orally, once daily starting from Cycle 1 Day 15 until disease progression, unacceptable toxicity (based on investigator assessment), or another treatment discontinuation criterion was met.
Period: Overall Study
Arm/Group | Cohort Dose Level (DL) 1 (Phase 1b): Erdafitinib 6 Milligrams (mg) + Cetrelimab 240/480 mg | Cohort DL2A (Phase 1b): Erdafitinib 8 mg + Cetrelimab 240/480 mg | Cohort DL2B (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg | Cohort DL2 (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg (RP2D) | Cohort DL2C (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Cisplatin 50 mg/m^2 | Cohort DL2D (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Carboplatin AUC 4 mg/mL/Min | Arm A (Phase 2): Erdafitinib 8/9 mg Monotherapy | Arm B (Phase 2): Erdafitinib 8 mg + Cetrelimab 240/480 mg
Started | 4 | 3 | 11 | 12 | 3 | 3 | 44 | 45
Treated (Treated Analysis Set) | 4 | 3 | 11 | 12 | 3 | 3 | 43 | 44
Completed | 4 | 3 | 5 | 3 | 2 | 2 | 21 | 17
Not Completed | 0 | 0 | 6 | 9 | 1 | 1 | 23 | 28
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Ongoing | 0 | 0 | 6 | 8 | 1 | 1 | 22 | 24
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set was defined as all participants who had received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort Dose Level (DL) 1 (Phase 1b): Erdafitinib 6 Milligrams (mg) + Cetrelimab 240/480 mg | Cohort DL2A (Phase 1b): Erdafitinib 8 mg + Cetrelimab 240/480 mg | Cohort DL2B (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg | Cohort DL2 (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg (RP2D) | Cohort DL2C (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Cisplatin 50 mg/m^2 | Cohort DL2D (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Carboplatin AUC 4 mg/mL/Min | Arm A (Phase 2): Erdafitinib 8/9 mg Monotherapy | Arm B (Phase 2): Erdafitinib 8 mg + Cetrelimab 240/480 mg | Total
Number analyzed (Participants) | 4 | 3 | 11 | 12 | 3 | 3 | 43 | 44 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 7 | 4 | 3 | 0 | 12 | 13 | 41
  >=65 years | 3 | 2 | 4 | 8 | 0 | 3 | 31 | 31 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (6.5) | 66.7 (9.07) | 61.3 (11.14) | 63.5 (11.41) | 60.3 (0.58) | 69 (3.61) | 71.1 (10.18) | 70.2 (8.61) | 68.8 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 5 | 0 | 1 | 10 | 11 | 30
  Male | 4 | 2 | 9 | 7 | 3 | 2 | 33 | 33 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 5
  Not Hispanic or Latino | 4 | 0 | 9 | 10 | 3 | 3 | 39 | 37 | 105
  Unknown or Not Reported | 0 | 2 | 2 | 1 | 0 | 0 | 3 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 1 | 1 | 3 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 1 | 6 | 11 | 2 | 2 | 36 | 36 | 98
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 3 | 1 | 0 | 0 | 4 | 6 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  BELARUS | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 10
  BELGIUM | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 5
  BRAZIL | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
  FRANCE | 0 | 2 | 2 | 1 | 0 | 0 | 3 | 4 | 12
  ITALY | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 2 | 8
  POLAND | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  RUSSIAN FEDERATION | 0 | 0 | 1 | 1 | 2 | 1 | 8 | 8 | 21
  SOUTH KOREA | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 2 | 8
  SPAIN | 2 | 1 | 4 | 6 | 0 | 0 | 4 | 8 | 25
  TAIWAN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  TURKEY | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 17
  UNITED KINGDOM | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
  UNITED STATES | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-Limiting Toxicity (DLTs)
Description: Number of participants with DLTs were reported. The DLTs as per National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE version 5.0) are specific adverse events defined as grade 3 (severe), grade 4 (life-threatening), and grade 5 (death) non-hematological toxicity or hematological toxicity.
Time Frame: Up to 8 weeks
Population: Treated analysis set included all participants who had received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort Dose Level (DL) 1 (Phase 1b): Erdafitinib 6 Milligrams (mg) + Cetrelimab 240/480 mg | Cohort DL2A (Phase 1b): Erdafitinib 8 mg + Cetrelimab 240/480 mg | Cohort DL2B (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg | Cohort DL2 (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg (RP2D) | Cohort DL2C (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Cisplatin 50 mg/m^2 | Cohort DL2D (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Carboplatin AUC 4 mg/mL/Min
Number analyzed (Participants) | 4 | 3 | 11 | 12 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 2: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by Investigator Assessment
Description: ORR is defined as the percentage of participants who achieved confirmed complete response (CR) or confirmed partial response (PR), according to response evaluation criteria in solid tumors (RECIST) version1.1. As per RECIST version 1.1, CR: disappearance of all lesions; all lymph nodes were non-pathological in size and normalization of tumor marker level; PR: greater than or equal to (>=) 30 percent (%) decrease in the sum of the diameters of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of nontarget lesions.
Time Frame: From Day 1 up to 36 months
Population: Treated analysis set included all participants who had received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A (Phase 2): Erdafitinib 8/9 mg Monotherapy | Arm B (Phase 2): Erdafitinib 8 mg + Cetrelimab 240/480 mg
Number analyzed (Participants) | 43 | 44
Percentage of Participants | 44.2 | 54.5

3. Primary Outcome: Phase 2: Number of Participants With Treatment-emergent Adverse Event (TEAEs)
Description: Number of participants with TEAEs were reported. An adverse event is any untoward medical event that occurs in a participant administered an investigational product and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs were defined as adverse events with onset or worsening on or after date of first dose of study treatment.
Time Frame: From Day 1 up to 36 months
Population: Treated analysis set included all participants who had received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Phase 2): Erdafitinib 8/9 mg Monotherapy | Arm B (Phase 2): Erdafitinib 8 mg + Cetrelimab 240/480 mg
Number analyzed (Participants) | 43 | 44
Participants | 43 | 44

4. Secondary Outcome: Phase 1b and Phase 2: Plasma Concentration of Erdafitinib
Time Frame: Up to 6 years 1 month
Reporting Status: Not Posted, anticipated posting 2026-06

5. Secondary Outcome: Phase 1b and Phase 2: Serum Concentration of Cetrelimab
Time Frame: Up to 6 years 1 month
Reporting Status: Not Posted, anticipated posting 2026-06

6. Secondary Outcome: Phase 1b: Plasma Concentration of Platinum (Cisplatin and Carboplatin) Chemotherapy
Time Frame: Up to 6 years 1 month
Reporting Status: Not Posted, anticipated posting 2026-06

7. Secondary Outcome: Phase 1b and Phase 2: Number of Participants With Anti-Cetrelimab Antibodies
Time Frame: Up to 6 years 1 month
Reporting Status: Not Posted, anticipated posting 2026-06

8. Secondary Outcome: Phase 2: Number of Participants With Serious Adverse Events (SAEs)
Time Frame: Up to 6 years 1 month
Reporting Status: Not Posted, anticipated posting 2026-06

9. Secondary Outcome: Phase 2: Number of Participants With Abnormal Laboratory Values
Time Frame: Up to 6 years 1 month
Reporting Status: Not Posted, anticipated posting 2026-06

10. Secondary Outcome: Phase 2: Duration of Response (DoR)
Time Frame: Up to 6 years 1 month
Reporting Status: Not Posted, anticipated posting 2026-06

11. Secondary Outcome: Phase 2: Time to Response (TTR)
Time Frame: Up to 6 years 1 month
Reporting Status: Not Posted, anticipated posting 2026-06

12. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Time Frame: Up to 6 years 1 month
Reporting Status: Not Posted, anticipated posting 2026-06

13. Secondary Outcome: Phase 2: Overall Survival (OS)
Time Frame: Up to 6 years 1 month
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: Phase 1b: From Day 1 up to 40 months; Phase 2: From Day 1 up to 36 months
Description: Treated analysis set included all participants who had received at least one dose of study drug.
Arm/Group | Cohort Dose Level (DL) 1 (Phase 1b): Erdafitinib 6 Milligrams (mg) + Cetrelimab 240/480 mg | Cohort DL2A (Phase 1b): Erdafitinib 8 mg + Cetrelimab 240/480 mg | Cohort DL2B (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg | Cohort DL2 (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg (RP2D) | Cohort DL2C (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Cisplatin 50 mg/m^2 | Cohort DL2D (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Carboplatin AUC 4 mg/mL/Min | Arm A (Phase 2): Erdafitinib 8/9 mg Monotherapy | Arm B (Phase 2): Erdafitinib 8 mg + Cetrelimab 240/480 mg
All-Cause Mortality (participants affected / at risk) | 4/4 | 3/3 | 5/11 | 3/12 | 2/3 | 2/3 | 21/43 | 17/44
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/3 | 4/11 | 6/12 | 3/3 | 1/3 | 22/43 | 19/44
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 11/11 | 12/12 | 3/3 | 3/3 | 43/43 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort Dose Level (DL) 1 (Phase 1b): Erdafitinib 6 Milligrams (mg) + Cetrelimab 240/480 mg (N=4) | Cohort DL2A (Phase 1b): Erdafitinib 8 mg + Cetrelimab 240/480 mg (N=3) | Cohort DL2B (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg (N=11) | Cohort DL2 (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg (RP2D) (N=12) | Cohort DL2C (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Cisplatin 50 mg/m^2 (N=3) | Cohort DL2D (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Carboplatin AUC 4 mg/mL/Min (N=3) | Arm A (Phase 2): Erdafitinib 8/9 mg Monotherapy (N=43) | Arm B (Phase 2): Erdafitinib 8 mg + Cetrelimab 240/480 mg (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Maculopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Punctate Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Serous Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal Mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis Infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Covid-19 Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes Ophthalmic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis Chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour Perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypovolaemic Shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort Dose Level (DL) 1 (Phase 1b): Erdafitinib 6 Milligrams (mg) + Cetrelimab 240/480 mg (N=4) | Cohort DL2A (Phase 1b): Erdafitinib 8 mg + Cetrelimab 240/480 mg (N=3) | Cohort DL2B (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg (N=11) | Cohort DL2 (Phase 1b): Erdafitinib 8/9 mg + Cetrelimab 240/480 mg (RP2D) (N=12) | Cohort DL2C (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Cisplatin 50 mg/m^2 (N=3) | Cohort DL2D (Phase 1b): Erdafitinib 8 mg + Cetrelimab 360 mg + Carboplatin AUC 4 mg/mL/Min (N=3) | Arm A (Phase 2): Erdafitinib 8/9 mg Monotherapy (N=43) | Arm B (Phase 2): Erdafitinib 8 mg + Cetrelimab 240/480 mg (N=44)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 3 | 3 | 2 | 16 | 17
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 3
Cataract (Eye disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3
Chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Conjunctival Hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Detachment of Macular Retinal Pigment Epithelium (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Detachment of Retinal Pigment Epithelium (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Dry Eye (Eye disorders) | 1 | 0 | 1 | 2 | 1 | 1 | 2 | 6
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Eyelid Oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 5 | 5
Lacrimal Disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 2
Macular Detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Posterior Capsule Opacification (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1
Serous Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2
Trichiasis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 5 | 4
Visual Acuity Reduced (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 4
Vitreous Floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 4 | 2 | 0 | 0 | 3 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Anal Fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal Inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 5 | 4 | 0 | 1 | 14 | 7
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 9 | 10 | 1 | 0 | 21 | 20
Dry Mouth (Gastrointestinal disorders) | 2 | 2 | 6 | 7 | 1 | 2 | 16 | 26
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Gingival Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 4 | 3 | 0 | 0 | 9 | 4
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 3 | 3 | 9 | 1 | 2 | 31 | 26
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 0 | 2 | 4 | 3
Asthenia (General disorders) | 0 | 1 | 4 | 7 | 1 | 0 | 5 | 10
Chills (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Face Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 2 | 1 | 0 | 1 | 10 | 11
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Localised Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 2 | 4 | 0 | 1 | 4 | 4
Xerosis (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Autoimmune Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gallbladder Polyp (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatobiliary Disease (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 2
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 4 | 0 | 0 | 1 | 3
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 6
Dermatophytosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Genital Herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Herpes Virus Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Klebsiella Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1
Oral Herpes (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis Externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 2 | 2 | 0 | 0 | 10 | 4
Perirectal Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rash Pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Skin Bacterial Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Strongyloidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 2 | 4 | 0 | 0 | 4 | 6
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Corneal Abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Persistent Corneal Epithelial Defect (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 4 | 1 | 1 | 1 | 14 | 11
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 3 | 2 | 2 | 1 | 10 | 8
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 5
Blood Calcium Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 2 | 3 | 1 | 0 | 7 | 10
Blood Parathyroid Hormone Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Blood Urea Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
International Normalised Ratio Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase Increased (Investigations) | 0 | 0 | 4 | 2 | 0 | 0 | 6 | 8
Weight Decreased (Investigations) | 0 | 2 | 2 | 1 | 0 | 0 | 7 | 8
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 3 | 5 | 1 | 0 | 8 | 9
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 4 | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 8 | 10 | 3 | 3 | 36 | 30
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 5
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 0 | 0 | 9 | 7
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3 | 0 | 1 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 2 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 1
Cardiac Myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Disturbance in Attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Dysgeusia (Nervous system disorders) | 2 | 2 | 2 | 4 | 1 | 0 | 7 | 9
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 5 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental Impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adjustment Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2
Mixed Anxiety and Depressive Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 6 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nephropathy Toxic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 3 | 2
Renal Pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Tract Pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scrotal Dermatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Scrotal Oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Testicular Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 4 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 2 | 0 | 1 | 3 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 4 | 0 | 1 | 6 | 5
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 4 | 0 | 1 | 15 | 17
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lichen Planus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lichen Sclerosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 7 | 3
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 1 | 0 | 4 | 6
Nail Dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 1 | 0 | 0 | 5 | 8
Nail Ridging (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Nail Toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 4 | 0 | 0 | 6 | 8
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 5 | 4
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 4 | 1 | 0 | 11 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 5 | 0 | 0 | 3 | 5
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 3
Peripheral Venous Disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT03473743/Prot_002.pdf
  • Statistical Analysis Plan (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT03473743/SAP_003.pdf